CLINICAL TRIAL: NCT07002931
Title: Effects of Three Different Surgical Techniques for Horizontal Ridge Bone Augmentation: A Superiority Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00012490
Record Dates: First submitted 2025-05-25; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Alveolar Bone Atrophy
Keywords: alveolar bone augmentation; horizontal bone augmentation
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: oral pathologist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- khoury block graft (Active Comparator): Bone blocks will be harvested from the retromolar area after measuring of the size required and measuring of the donor site anatomy. Piezoelectric device will be used to perform the graft osteotomy. The osteotomy lines will be connected and the graft will be mobilized using a bibeveled chisel and mallet. Sharp bony edges will be smoothened and the donor defect was packed with gelatin sponges. The bone block margins will be smoothened and separated into two thinner bone shells using titanium disk with copious saline irrigation. The blocks will be fixed into the recipient site buccally using at least two microscrews leaving a gap to be filled with bone graft. Particulate xenogenic bone graft will be mixed with the autogenous bone chips (50% Xenograft: 50% Autogenous graft) to fill the gap between the buccal bone plate and the fixed bone shells. The augmented site will be covered with a pericardium membrane.
  Interventions: Procedure: khoury block graft
- urban sausage technique (Active Comparator): A resorbable pericardium membrane will be fixed with titanium pins on the lingual bone plate (2-3mm from the bone crest) and on the buccal bone plate allowing for packing of particulate mix of bone graft (50% Xenograft: 50% Autogenous graft). Overfilling of the graft will be respected to compensate for future resorption. The membrane will be stretched over the graft ensuring maximum immobilization of the graft.
  Interventions: Procedure: urban sausage technique
- guided bone regeneration using PTFE membrane (Active Comparator): A non-resorbable polytetrafluoroethylene (PTFE) membrane will be fixed with titanium tacks on the lingual bone plate (2-3mm from the bone crest) and on the buccal bone plate allowing for packing of particulate mix of bone graft (50% Xenograft: 50% Autogenous graft). Overfilling of the graft will be respected to compensate for future resorption.
  Interventions: Procedure: non resorbable membrane

INTERVENTIONS:
Procedure: khoury block graft — Bone blocks will be harvested from the retromolar area after measuring of the size required and measuring of the donor site anatomy. Piezoelectric device will be used to perform the graft osteotomy. The osteotomy lines will be connected and the graft will be mobilized using a bibeveled chisel and mallet. Sharp bony edges will be smoothened and the donor defect was packed with gelatin sponges. The bone block margins will be smoothened and separated into two thinner bone shells using titanium disk with copious saline irrigation. The blocks will be fixed into the recipient site buccally using at least two microscrews leaving a gap to be filled with bone graft. Particulate xenogenic bone graft will be mixed with the autogenous bone chips (50% Xenograft: 50% Autogenous graft) to fill the gap.
  Arms: khoury block graft
Procedure: urban sausage technique — : A resorbable pericardium membrane will be fixed with titanium pins on the lingual bone plate (2-3mm from the bone crest) and on the buccal bone plate allowing for packing of particulate mix of bone graft (50% Xenograft: 50% Autogenous graft). Overfilling of the graft will be respected to compensate for future resorption. The membrane will be stretched over the graft ensuring maximum immobilization of the graft.
  Arms: urban sausage technique
Procedure: non resorbable membrane — A non-resorbable polytetrafluoroethylene (PTFE) membrane (Permamem membrane, Botiss Biomaterials, Germany) will be fixed with titanium tacks on the lingual bone plate (2-3mm from the bone crest) and on the buccal bone plate allowing for packing of particulate mix of bone graft (50% Xenograft: 50% Autogenous graft). Overfilling of the graft will be respected to compensate for future resorption.
  Arms: guided bone regeneration using PTFE membrane

SUMMARY:
the goal of this clinical trial in to investigate the efficacy of three different horizontal augmentation techniques with regards to the volume of bone gained, the quality of the bone gained and the level of patient pain scale.

Researchers will compare the volume of bone gained radiographically and the quality of the bone gain using histological analysis.

the participants in this study will be required to record and submit a pain scale chart.

DETAILED DESCRIPTION:
Introduction While preservation of the dentition is the goal of dentistry, tooth loss may occur for a variety of reasons including fracture, pulpal infection, severe periodontal disease, or pathological processes. Following tooth extraction, crestal bone resorption and invagination of the soft tissue will occur (1-3).

In cases of severe bone loss-potentially due to a significant timelapse since extraction, unfavorable occlusal load, (traumatic occlusion), infection, trauma? or periodontal disease-bone frequently needs to be augmented prior to or during implant placement (4,5). Different augmentation techniques have been developed depending on localization, extent, and configuration of the bone defect (6,7).

While some consider autogenous bone grafts the gold standard for guided bone regeneration, others consider a combination of resorbable collagen membrane and inorganic bovine bone as the standard method for guided bone regeneration (GBR). Many studies demonstrate that autologous grafts are highly reliable for increasing bone volume prior to placing implants (8-10).

Different techniques for GBR have evolved based on the properties of available bone grafts and membranes, with the goal of optimizing osteoblastic potential while preventing epithelial and connective tissue invagination into the bone graft. Karring and others (11) suggested that the ideal membrane is biocompatible, occludes connective tissue cells from the bone, integrates well with the host tissues, helps achieve bone graft stability, and maintains space in a clinically manageable scenario. Autogenous bone grafts have the benefit of supplying osteoinductive growth factors, an osteoconductive scaffold, and osteogenic cells but can be more quickly resorbed than xenografts which typically provide the osteoconductive scaffold.

Although many different classes of GBR membranes are commercially available, these can be generally divided into two categories: non-resorbable and resorbable membranes (14). Synthetic and naturally derived resorbable membranes have been developed to avoid the need for a second surgical intervention and to reduce the risks of membrane exposure. However, the variability in resorption rate and poor mechanical properties of the resorbable membranes are significant limiting factors (15).

Among the non-resorbable membranes, the expanded polytetrafluoroethylene (ePTFE) membranes have been accepted as the gold standard material in GBR for their mechanical stability, biocompatibility, lack of foreign body response after implantation, prevention of tissue ingrowth during the process of bone regeneration and the ability to facilitate bone regeneration in many clinical studies (16,17). However, non-resorbable membranes suffer from various drawbacks, as their stiffness may cause soft tissue dehiscence, which can lead to the membrane exposure and subsequent infection. Additionally, a second surgery is needed to remove non-resorbable membranes, resulting in patient discomfort and higher economic burden (19,20).

Three commonly used techniques for guided bone regeneration include the sausage technique, Khoury technique, and use of an ePTFE membrane with autogenous bone (a common method for conventional guided bone regeneration). The sausage technique introduced by Istvan Urban utilizes a combination of 50% autogenous bone and 50% xenogenic bone. The technique was reported to enable successful bone regeneration by immobilizing the collagen membrane with a titanium pin and pushing the bone graft material in the crestal direction (22). The technique is similar to conventional GBR in that the membrane is fixed with pins. However, the graft material is filled inside the fixed membrane in a sufficient quantity to show a balloon effect and to push the graft material in the crestal direction to create tension on the membrane (23).

The Khoury technique uses a MicroSaw to obtain a bone block from the ramus or symphysis. The block is longitudinally dissected with the MicroSaw and bone scrapings are removed from the surface until each block is approximately 1mm thick. Microscrews are used to attach the first block graft, the particulate is placed between the block and ridge, and then the second block graft completes the anatomical reconstruction.

While many studies look at a comparison of two guided bone regeneration techniques, from a histological or clinical perspective, there is no clinical evidence comparing the three different regenerative techniques from a clinical, radiographic, and histological manner. Thus, this clinical study will have three general aims:

Objective The aim of the present study is to compare three different ridge bone regeneration techniques for horizontal bone augmentation. The null is that no statistically significant differences will be observed.

Material and Methods Study design This will be a 3-arm multicentric single-blind randomized clinical trial. Patient Selection Patients will be included in two different clinics with two different operators. The enrollment will follow the following inclusion criteria, 1) Have two or more missing teeth in the posterior mandibular segment; 2) The alveolar ridge in the edentulous site of the selected patients will have a buccolingual width of less than 4mm; 3) Sufficient vertical bone height; 4) Free of any local or systemic condition that may contraindicate ridge expansion procedure; 5) No sex predilection; 6) The patient will be between the ages of 18-70. The exclusion criteria are: 1) Patients taking any medication that may interfere with bone healing or bone biology; 2) Patients with any systemic disease that may affect bone healing; 3) Any patients with any previous bone grafting procedure at the site of interest; 4) Smokers; 5) Patient's that have been diagnosed with periodontal disease, as sufficient ridge height would be improbable. The patients will be fully informed about the surgical procedures and the alternative treatments. Benefits and risks of the procedures will be explained and all patients. All the patients should sign a written consent before the being enrolled in the study. The study protocol will be register at a clinical trial platform.

Sample size calculation The sample size analysis was performed considering the null hypothesis that no difference would be found between the 3 different groups regarding the primary outcome, the horizontal dimension (labio-palatal) (mm). Using the alpha (α) level of 0.05, a beta (β) level of 0.2 (power = 80%), a standard deviation of 1.0mm , and a difference of 1.0mm between groups, 21 subjects would be necessary for each group. Therefore, 63 patients will be included.

Pre-operative Examination Pre-operative examination of each patient will include clinical examination that includes a full periodontal chart (probing depths, clinical attachment level, preoperative impressions and photographs).

Cone Beam Volumetric Topography (CBVT) will be used with an acrylic template with a radiopaque indicator in place to determine the exact site of measurement, and to allow for accurate measurements of the bone width postoperatively in the same site. The radiopaque indicator will be placed in the middle of the proposed grafting site mesiodistally.

Randomization and allocation concealment The patients will be randomly divided into three groups. The first group will receive autogenous bone block grafts fixed at a distance (Khoury technique), the second group will receive augmentation using pericardium membrane fixed with tacks (Urban Sausage technique), while the third group will receive augmentation using non-resorbable membrane fixed with tacks. In each center, a person not involved in the study will be responsible for randomization and allocation concealment. The random allocation sequence will be generated using computer software, and then the randomization codes will be placed and sealed in opaque envelopes. Each patient's envelope will only be opened before the surgical procedure.

Surgical procedures All investigators in charge of the surgical procedure will participate in a calibration meeting. The surgical procedure will be standardized through discussions, case presentations, step-by-step reviews, and videos. This same procedure will be repeated when half of the surgeries is completed.

The patients will be medicated with midazolam 10mg (Dormicum, Roche) intramuscular 1 hour before the procedure. The patients will be asked to rinse with 0.125% Chlorhexidine mouthwash for 30 seconds immediately before the procedure. The procedures will be performed under local anesthesia. Inferior alveolar and mental nerve block will be used (Articaine 4% 1:100.000 epinephrine). Local infiltration will be used in the site for hemostasis.

A mandibular posterior midcrestal incision will be performed within the keratinized mucosa with intrasulcular buccal and lingual incisions at the anterior adjacent teeth including divergent-releasing incision. Another distal releasing incision will be performed. Full mucoperiosteal flaps will be elevated on buccal and lingual aspects. Retraction sutures will be used. Curettage of the bony crest of any soft tissue remnants will take place. A periodontal probe will be used to measure the approximate size of the block graft to be harvested. Decortication of the buccal bone plate will be done using round bur under copious saline irrigation. Then, the area will be grafting using one of the three techniques indicated below.

Group 1 - Block graft (Khoury Technique): Bone blocks will be harvested from the retromolar area after measuring of the size required and measuring of the donor site anatomy. Piezoelectric device will be used to perform the graft osteotomy. The block size should be slightly larger than the defect size. The osteotomy lines will be connected and the graft will be mobilized using a bibeveled chisel and mallet. Elevation starts from the coronal osteotomy line. Sharp bony edges will be smoothened and the donor defect was packed with gelatin sponges. The bone block margins will be smoothened and separated into two thinner bone shells using titanium disk with copious saline irrigation. The blocks will be fixed into the recipient site buccally using at least two microscrews (Devemed GmbH, Germany) leaving a gap to be filled with bone graft. Auto chip maker (ACM) bur (Neobiotech, Korea) will be used to collect autogenous bone chips from the external oblique ridge area. Particulate xenogenic bone graft (Geistlich Bio-Oss, Germany) will be mixed with the autogenous bone chips (50% Xenograft: 50% Autogenous graft) to fill the gap between the buccal bone plate and the fixed bone shells. The augmented site will be covered with a pericardium membrane (Jason, Botiss biomaterials, Germany).

Group 2 - Urban Sausage Technique: A resorbable pericardium membrane (Jason membrane, Botiss Biomaterials, Germany) will be fixed with titanium pins (Devemed GmbH, Germany) on the lingual bone plate (2-3mm from the bone crest) and on the buccal bone plate allowing for packing of particulate mix of bone graft (50% Xenograft: 50% Autogenous graft). Overfilling of the graft will be respected to compensate for future resorption. The membrane will be stretched over the graft ensuring maximum immobilization of the graft.

Group 3 - Non-resorbable membrane: A non-resorbable polytetrafluoroethylene (PTFE) membrane (Permamem membrane, Botiss Biomaterials, Germany) will be fixed with titanium tacks (Devemed GmbH, Germany) on the lingual bone plate (2-3mm from the bone crest) and on the buccal bone plate allowing for packing of particulate mix of bone graft (50% Xenograft: 50% Autogenous graft). Overfilling of the graft will be respected to compensate for future resorption.

Periosteal releasing incision of the buccal flap and releasing of the lingual flap from the underlying mylohyoid attachment will be done to ensure proper immobilization of the flaps and tension-free primary wound closure.

Wound closure will be achieved using 5-0 non-resorbable polypropylene sutures. Double layer suturing technique will be used with horizontal mattress sutures 5mm below the incision line followed with interrupted or continuous with lock sutures crestally. interrupted sutures will be used for vertical releasing incisions.

Post-operative instructions All the patients will receive Augmentin (Amoxicillin/clavulanic acid 1g) every 12 hours for 5 days and ibuprofen 600mg every 8 hours for 5 days. 0.125% Chlorhexidine mouthwash will be used twice daily for 10 days. Sutures will be removed after 14 days.

Evaluations

1. Cone Beam Volumetric Topography (CBVT). Two CBVT, one before and one after 6 months will be recorded with the previously used acrylic template with a radiopaque indicator in place. One single examiner who will be blinded and calibrated for the procedures will evaluate the images. For the calibration, the examiner will evaluate 10 images 2 times within 24 hours apart and will measure the primary outcome, i.e. horizontal bone thickness. The agreement of the measurements will be assessed with the intra-class correlation. The following measures will be assessed: 1) Horizontal bone thickness, measured in 3 levels (3, 5, and 7mm distant from the bone crest); 2) Bone Height, the distance between the bone crest and a fixed reference point; 3) Horizontal and Height Bone Gain, the variation between baseline and the final measures of both parameters (Δ=final-initial). In addition, the volume of bone gain will be assessed.
2. Patient-centred outcomes. Postoperative pain and discomfort and analgesic consumption will be assessed using a questionnaire during the following 7 postoperative days. The patients will be requested to monitor their postoperative pain/discomfort and the number of days on analgesics during this period.
3. Histological analysis. After 6 months, the site will be re-opened. The flap outline will be similar to the first surgery. The surgical access will be limited to the crestal area except for group 3. Titanium screws will be removed in group 1. Non-resorbable membrane and pseudo-membrane layer will be removed in group 3. A 2mm trephine bur will be used to collect a core biopsy at the preplanned implant positions for histomorphometric analysis. Root-form dental implants will be placed with the proper lengths and diameters. Area and percentage of areas will be assessed for the newly formed bone, the bone marrow spaces, and bone graft particles.
4. Clinical measurement: the frequency of complications, i.e. episodes of suppuration, membrane exposure, and suture dehiscence, will be recorded. In addition, the implant insertion torque will be evaluated.

Statistical analyses Descriptive statistics will be expressed as mean ± standard deviation and percentage. Normality will be tested using the Shapiro-Wilk test. Values referring to VAS scores will be compared using One-way ANOVA (Wilcoxon in case of the non-normal distribution data), the horizontal bone gain will be assessed with Repeated Measures of Variance. The frequency of sites effects will be assessed with X2. For the histological analyses, the volume of vital bone, graft remnants, and connective tissue will be measured based on the averages of the percentages and compared using One-way ANOVA (Wilcoxon in case of the non-normal distribution data). A significance of 5% will be used for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Have two or more missing teeth in the posterior mandibular segment; 2) The alveolar ridge in the edentulous site of the selected patients will have a buccolingual width of less than 4mm; 3) Sufficient vertical bone height; 4) Free of any local or systemic condition that may contraindicate ridge expansion procedure

Exclusion Criteria:

* : 1) Patients taking any medication that may interfere with bone healing or bone biology; 2) Patients with any systemic disease that may affect bone healing; 3) Any patients with any previous bone grafting procedure at the site of interest; 4) Smokers; 5) Patient's that have been diagnosed with periodontal disease, as sufficient ridge height would be improbable.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
post operative pain scale | 7 days
  participants will be asked to assess and record the level of pain daily on a pain chart submitted to them post operatively.

SECONDARY OUTCOMES:
horizontal bone gain | 6 months
  the participants will undergo radiographic analysis using CBCT scans performed preoperatively, immediately post operative and six months post operative respectively. the scans will be used to assess the amount of bone gain for each procedure
qualitative bone assessment | 6 months
  core biopsy will be obtained from the grafted sites six months post operatively to assess the quality of the regenerated bone

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, British university of egypt, Cairo, Egypt